CLINICAL TRIAL: NCT06141538
Title: Response of Intracardiac Thrombus to Anticoagulants in Patients With Non-valvular Atrial Fibrillation (LYSIS): an Investigator-initiated, National, Multicenter, Retrospective-prospective, Observational Cohort Study
Brief Title: Response of Intracardiac Thrombus to Anticoagulants in Patients With Non-valvular Atrial Fibrillation (LYSIS)
Acronym: LYSIS
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: 521 Hospital of NORINCO Group (Other); Shaanxi Provincial People's Hospital (Other); Xiangyang Central Hospital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-404
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation; Intracardiac Thrombus
Keywords: Atrial Fibrillation; Intracardiac Thrombus; Anticoagulation Therapy; Major adverse cardiovascular and cerebrovascular events
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Adequate and regular anticoagulant therapy. Anticoagulation therapy is determined based on the patient's CHADS₂ or CHA₂DS₂-VASc score. Anticoagulant medications include vitamin K antagonists, novel oral anticoagulants (NOACs), and aspirin.
  Interventions: Other: Observational; No Interventions were given.
- Control group: Patients who have not received regular or continuous anticoagulation therapy due to poor compliance or other reasons.
  Interventions: Other: Observational; No Interventions were given.

INTERVENTIONS:
Other: Observational; No Interventions were given. — Observational; No Interventions were given.

SUMMARY:
This study aims to analyze changes in the immune status, metabolic status, and host microbiome community structure in non-valvular atrial fibrillation patients with intracardiac thrombus. Additionally, the study aims to analyze factors that influence the responsiveness and occurrence of adverse events related to anticoagulant therapy.

DETAILED DESCRIPTION:
The researcher-initiated clinical cohort study is a national multicenter, retrospective-prospective study of non-valvular atrial fibrillation patients with intracardiac thrombus, based on molecular biology and multi-omics analysis. The study aims to analyze the changes in the body's immune status, metabolic status, and host microbiome community structure, as well as to analyze the factors that influence the responsiveness of intracardiac thrombus to anticoagulant therapy. The study also evaluates the occurrence of adverse events related to anticoagulation in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, age ≤80 years old
* Patients with atrial fibrillation detected by routine surface 12-lead electrocardiography or Holter
* Transesophageal echocardiography confirmed the presence of cardiac thrombus, and the patient had not received any anticoagulant therapy

Exclusion Criteria:

* Echocardiography confirmed valvular heart disease
* Contraindications to anticoagulants
* Patients with the previous history of hemorrhagic stroke
* Low platelet count or functional platelet defects
* Congenital or acquired coagulation or bleeding disorders
* Abnormal liver function (liver enzymes >2 times the upper limit)
* Renal failure (endogenous creatinine clearance <30ml/min)
* Surgery was planned within the intended study time or had been operated within 30 days before the study
* Other comorbidities that can cause bleeding, such as tumors
* Patients with autoimmune diseases or immunodeficiency, or patients who are currently using immunosuppressants and immunomodulators
* Patients are currently participating in other clinical studies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation who have been diagnosed with intracardiac thrombosis by First Affiliated Hospital of Xi'an Jiaotong University and multiple medical centers, meet the indications for anticoagulation therapy, and are willing to receive anticoagulation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of thrombolysis | 1，2，3 months after enrollment.
  Success rate of thrombolysis within 3 months after initiating anticoagulation therapy.
Change of incidence of MACCE | 1，2，3 months after enrollment.
  Major adverse cardiovascular and cerebrovascular events, a composite of all-cause mortality, myocardial infarction, coronary revascularization, and stroke.

SECONDARY OUTCOMES:
Change of incidence of adverse anticoagulation events | 1，2，3 months after enrollment.
  Bleeding and thrombotic events
Change of incidence of all-cause mortality | 1，2，3 months after enrollment.
  All-cause mortality diagnosed by clinical doctors.
Change of incidence of myocardial infarction | 1，2，3 months after enrollment.
  Myocardial infarction diagnosed by clinical doctors.
Change of incidence of coronary revascularization | 1，2，3 months after enrollment.
  Coronary revascularization assessed by clinical doctors.
Change of incidence of stroke | 1，2，3 months after enrollment.
  Stroke diagnosed by clinical doctors.

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Li, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Chaofeng Sun, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiantong University, Xi'an, Shaanxi, China